CLINICAL TRIAL: NCT05290402
Title: Development of an Application-Based Digital Navigator for Perioperative Breast Surgery Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1211; NCI-2022-01986 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- an application-based digital navigator: JEEVA" is a new digital health navigator app. This app can be used on a mobile phone or tablet. JEEVA has all of the surgical teaching information from the traditional paper packet and also has additional resources like brief videos, checklists, and reference photos.
  Interventions: Other: JEEVA (new digital health navigator app)

INTERVENTIONS:
Other: JEEVA (new digital health navigator app) — An app can be used on a mobile phone or tablet.

SUMMARY:
The goal of this research study is to learn how accessible JEEVA is for patients during the perioperative period (the time after the pre-operative surgical appointment, and up to 30 days after surgery

DETAILED DESCRIPTION:
Objectives:

Demonstrate feasibility of use for a mobile device-based application to provide perioperative resources and support in a multimedia format to breast surgery patients

Measure ease of use, interface and satisfaction with the electronic delivery of materials through the mobile health (mHealth) App Usability Questionnaire (MAUQ)

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this study include breast surgical patients 18 years of age and older evaluated at the Texas Medical Center campus in the Nellie B Connally breast center or in the Houston Area Locations (HALs).

This includes patients undergoing excisional biopsy, segmental mastectomy, total mastectomy, skin-sparing mastectomy, nipple-sparing mastectomy, sentinel lymphadenectomy, targeted axillary lymphadenectomy, axillary lymphadenectomy, and axillary reverse mapping.

Exclusion Criteria:

Patients who do not have a smartphone), which utilizes iOS or Android operating systems,

Patients who have visual impairment or blindness, which precludes effective utilization of an app, will be excluded.

Patients whose surgical planning is discussed by telephone outside of an in-person pre-operative visit, will be excluded from the study.

Patients who have cognitive impairment will be exclude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Surgery Patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Measure ease of use, interface and satisfaction with the electronic delivery of materials through the mobile health (mHealth) App Usability Questionnaire (MAUQ) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christina Checka, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT05290402/ICF_000.pdf